CLINICAL TRIAL: NCT00104806
Title: Phase II Trial of Arsenic Trioxide and Dose-Escalated Cholecalciferol in Myelodysplastic Syndrome
Brief Title: Arsenic Trioxide and Cholecalciferol (Vitamin D) in Treating Patients With Myelodysplastic Syndromes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: sponsor discontinues support
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000415574; CCCWFU-29304; CCCWFU-BG04-452
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: de novo myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; refractory anemia with excess blasts in transformation; refractory anemia with excess blasts; refractory anemia; refractory anemia with ringed sideroblasts; refractory cytopenia with multilineage dysplasia; chronic myelomonocytic leukemia; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Myeloproliferative Disorders; Anemia, Refractory, with Excess of Blasts; Anemia, Refractory; Leukemia, Myelomonocytic, Chronic | interventions — Cholecalciferol; Arsenic Trioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: cholecalciferol — 100 milligrams orally once a day for 28 days
Drug: arsenic trioxide — 0.3 milligram/kilogram weight intravenously for 5 days (loading) then 0.25/kg weight intravenously biweekly

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as arsenic trioxide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Cholecalciferol (vitamin D) may help cancer cells become normal cells. Giving arsenic trioxide together with cholecalciferol (vitamin D) may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving arsenic trioxide together with cholecalciferol (vitamin D) works in treating patients with myelodysplastic syndromes.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the complete response rate and the rate of hematological improvement in patients with myelodysplastic syndromes treated with arsenic trioxide and cholecalciferol (vitamin D).

Secondary

* Determine the safety of this regimen in these patients.
* Determine the time to progression to acute myeloid leukemia, defined as blast ≥ 20%, in patients treated with this regimen.
* Determine overall survival and progression-free survival of patients treated with this regimen.
* Determine the effect of this regimen on bone marrow and peripheral blood mononuclear cell apoptosis and p21 protein expression in these patients.

OUTLINE: This is an open-label, nonrandomized study.

Patients receive oral cholecalciferol (vitamin D)* once daily on days 1-28. Patients also receive arsenic trioxide IV over 1-4 hours on days 1-5 (week 1) and then twice weekly for 3 weeks (weeks 2-4) for course 1 and twice weekly for 4 weeks for all subsequent courses. Courses repeat every 28 days for up to 12 months in the absence of disease progression or unacceptable toxicity.

NOTE: * Patients who do not achieve a complete hematologic response receive escalating doses of cholecalciferol (vitamin D) at 3, 6, and 9 months during therapy in the absence of disease progression and unacceptable toxicity.

At the completion of study treatment, patients are followed for survival.

PROJECTED ACCRUAL: A total of 25-60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of myelodysplastic syndromes (MDS)

  * Bone marrow aspirate and biopsy with karyotyping performed within the past 12 weeks

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* ECOG 0-2

Life expectancy

* More than 6 months

Hematopoietic

* Ferritin ≥ 50 ng/mL
* Folate (serum and/or red blood cell) normal

Hepatic

* Not specified

Renal

* Creatinine < 2.0 mg/dL
* No history of hypercalcemia

Cardiovascular

* Absolute QT interval ≤ 460 msec by EKG with normal potassium and magnesium levels

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 weeks after study participation
* Serum vitamin B_12 normal

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior biologic therapy allowed
* More than 28 days since prior hematopoietic growth factors (e.g., filgrastim [G-CSF], sargramostim [GM-CSF], or epoetin alfa) for MDS
* No concurrent hematopoietic growth factors (e.g., G-CSF, GM-CSF, or epoetin alfa)
* No concurrent interleukin-11

Chemotherapy

* Prior chemotherapy allowed

Endocrine therapy

* Not specified

Radiotherapy

* Prior radiotherapy allowed

Surgery

* Not specified

Other

* More than 28 days since prior therapy for MDS except supportive therapy
* No concurrent cholecalciferol (vitamin D) analog, including topical therapy
* No concurrent vitamins or supplements containing cholecalciferol (vitamin D)
* No other concurrent therapy for MDS

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2004-11; Primary Completion 2006-01 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Complete response rate | 6 months
toxicity assessment after therapy | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Istvan Molnar, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States